CLINICAL TRIAL: NCT01673646
Title: A Multicenter, Open-label, Randomized, Phase II Study to Evaluate Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Pasireotide LAR in Japanese Patients With Active Acromegaly or Pituitary Gigantism
Brief Title: Efficacy and Safety of Pasireotide LAR (Long-acting Release) in Japanese Patients With Acromegaly or Pituitary Gigantism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230C1202
Record Dates: First submitted 2012-08-16; First posted 2012-08-28 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-07

CONDITIONS: Acromegaly; Pituitary Gigantism
Keywords: SOM230; Pasireotide; acromegaly; Phase II; growth disorder; gigantism; Pituitary adenoma; pituitary gigantism
MeSH Terms: conditions — Acromegaly; Gigantism; Growth Disorders; Pituitary Neoplasms | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pasireotide LAR 20mg (Experimental): Enrolled patients were randomized to 20mg pasireotide LAR.
  Interventions: Drug: Pasireotide LAR
- Pasireotide LAR 40mg (Experimental): Enrolled patients were randomized to 40mg pasireotide LAR.
  Interventions: Drug: Pasireotide LAR
- Pasireotide LAR 60mg (Experimental): Enrolled patients were randomized to 60mg pasireotide LAR.
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide LAR — Intramuscular administration of pasireotide LAR was repeated every month (1 month = 28 days) for 12 months in core phase. It was permitted to increase the dose up to 60 mg in a patient showing the following biochemical test results after 3 and 6 months of study treatment: mean GH levels ≥2.5 µg/L and/or IGF-1 > ULN. In the event of any problem with tolerability, it was permitted to reduce the next lower dosage level at any time.
  Other Names: SOM230

SUMMARY:
To evaluate efficacy, safety, pharmacokinetics and pharmacodynamics of pasireotide LAR in Japanese patients with active acromegaly or pituitary gigantism. Primary objective was to assess the total-group efficacy of pasireotide LAR on the reduction of mean GH levels to < 2.5 µg/L and the normalization of insulin-like growth factor-1 (IGF-1) at 3 months of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medication naïve acromegaly or pituitary gigantism
* Patients with inadequately controlled acromegaly or pituitary gigantism

Exclusion Criteria:

* Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1c >8%
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment
* Patients with risk factors for torsade de pointes, i.e. patients with a baseline QTcF > 470 ms, hypokalemia, hypomagnesemia, hypocalcemia, family history of long QT syndrome, or patients receiving a concomitant medication known to prolong QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Japan (27):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were planned and 33 patients were enrolled. The full analysis sets (FAS) consisted of 33 patients (11 patients per dose group).
Period: Overall Study
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Started | 11 | 11 | 11
Entered/Treated in Core Phase | 11 | 11 | 11
Completed Core Phase | 9 | 10 | 10
Entered Ext. Phase | 7 | 9 | 9
Did Not Enter Ext. Phase | 2 | 1 | 1
Treated Beyond 24 Months | 7 | 8 | 8
Discontinued Beyond 24 Months | 0 | 4 | 1
Completed | 7 | 4 | 7
Not Completed | 4 | 7 | 4
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 2 | 0
Not completed — Condition no longer requires study drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Completed Core/did not enter Ext. | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set comprises all patients to whom study treatment had been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg | Total
Number analyzed (Participants) | 11 | 11 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full analysis set comprises all patients to whom study treatment had been assigned by randomization.
  Years | 57.2 (11.48) | 49.1 (13.75) | 46.6 (14.60) | 51.0 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set comprises all patients to whom study treatment had been assigned by randomization.
  Participants
    Female | 4 | 7 | 2 | 13
    Male | 7 | 4 | 9 | 20
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full analysis set comprises all patients to whom study treatment had been assigned by randomization.
  Participants
    Asian | 11 | 11 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Total-group Response Rate at Month 3
Description: Percentage of participants with a reduction of mean growth hormone (GH) levels to < 2.5 µg/L and the normalization of insulin-like growth factor-1 (IGF-1) to within normal limits (age and sex related) at 3 months across all doses
Time Frame: Month 3
Population: The Full analysis Set (FAS): Comprises all patients to whom study treatment has been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the study treatment they have been assigned to during the randomization procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pasireotide LAR - All Participants: All patients randomized regardless of pasireotide LAR dose.
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants | 18.2 [7.0 to 35.5]

2. Secondary Outcome: Response Rate at Month 3 by Randomized Dose Level
Description: Percentage of participants with a reduction of mean GH levels to < 2.5 µg/L and the normalization of IGF-1 to within normal limits (age and sex related) at 3 months in each starting dose.
Time Frame: Month 3
Population: FAS: Comprises all patients to whom study treatment has been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the study treatment they have been assigned to during the randomization procedure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
Percentage of participants | 9.1 [0.2 to 41.3] | 36.4 [10.9 to 69.2] | 9.1 [0.2 to 41.3]

3. Secondary Outcome: GH Response at Month 3 by Randomized Dose
Description: Percentage of participants with a reduction of mean GH levels to < 2.5 µg/L at 3 months.
Time Frame: Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
Percentage of participants | 27.3 [6.0 to 61.0] | 45.5 [16.7 to 76.6] | 18.2 [2.3 to 51.8]

4. Secondary Outcome: IGF-1 Response at Month 3 by Randomized Dose
Description: Percentage of participants with the normalization of IGF-1 to within normal limits (age and sex related) at 3 months.
Time Frame: Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
Percentage of participants | 18.2 [2.3 to 51.8] | 45.5 [16.7 to 76.6] | 9.1 [0.2 to 41.3]

5. Secondary Outcome: Total-group Response Rate (GH & IGF-1) Over Time (Core Phase)
Description: Percentage of participants with a reduction of mean GH levels to < 2.5 µg/L and the normalization of IGF-1 to within normal limits (age and sex related) at 3, 6, 9 and 12 months
Time Frame: Months 3, 6, 9 & 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants
  Month 3 | 18.2 [7.0 to 35.5]
  Month 6 | 21.2 [9.0 to 38.9]
  Month 9 | 21.2 [9.0 to 38.9]
  Month 12 | 15.2 [5.1 to 31.9]

6. Secondary Outcome: Percentage of Overall Participants With the Reduction of GH Levels to <2.5 ug/L by Visit (Core Phase)
Description: This refers to the percentage of participants with a reduction of growth hormone (GH) response rates to <2.5 ug/L over time.
Time Frame: Months 3, 6, 9, 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percenage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percenage of participants
  Month 3 | 30.3 [15.6 to 48.7]
  Month 6 | 33.3 [18.0 to 51.8]
  Month 9 | 30.3 [15.6 to 48.7]
  Month 12 | 36.4 [20.4 to 54.9]

7. Secondary Outcome: Percentage of Overall Participants With the Normalization of IGF-1 by Visit (Core Phase)
Description: This refers to the percentage of participants with the normalization of insulin-like growth factor-1 (IGF-1) to within normal limits by visit.
Time Frame: Months 3, 6, 9, 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants
  Month 3 | 24.2 [11.1 to 42.3]
  Month 6 | 33.3 [18.0 to 51.8]
  Month 9 | 39.4 [22.9 to 57.9]
  Month 12 | 27.3 [13.3 to 45.5]

8. Secondary Outcome: Summary of Pasireotide LAR PK Parameters of Ctrough & Cmax by Randomized Dose Level
Description: Ctrough: The trough level concentration on day 28, 3 months post 1st, 2nd and 3rd injections of Pasireotide LAR.
  Cmax: The maximum concentration 3 months post the 1st injection and 3rd injection of LAR.
Time Frame: Ctrough: Day 28 after each injection 1-3, Cmax: 3 months after injections 1 and 3
Population: The pharmacokinetic (PK) analysis set (PAS) consists of full analysis set (FAS) who have evaluable PK concentration data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
ng/mL
  Ctrough Day 28, 1st inj | 5.36 (3.35) | 8.41 (5.26) | 10.8 (5.12)
  Ctrough Day 28, 2nd inj: number analyzed (Participants) | 11 | 10 | 11
  Ctrough Day 28, 2nd inj | 5.86 (2.38) | 10.7 (4.14) | 15.0 (9.12)
  Ctrough Day 28, 3rd inj: number analyzed (Participants) | 9 | 8 | 8
  Ctrough Day 28, 3rd inj | 5.85 (2.28) | 12.2 (6.75) | 11.1 (4.99)
  Cmax, 1st inj | 7.19 (3.48) | 10.3 (7.25) | 17.0 (13.7)
  Cmax, 3rd inj: number analyzed (Participants) | 9 | 8 | 8
  Cmax, 3rd inj | 8.23 (2.35) | 17.3 (9.61) | 16.2 (7.12)

9. Secondary Outcome: Summary of Pasireotide LAR PK Parameter of Accumulation Ratio Randomized Dose Level
Description: The accumulation ratio was calculated as a ratio of (Ctrough day28, 3rd injection/Ctrough day28, 1st injection).
Time Frame: Day 28 after injections 1 and 3
Population: PAS: Consists of full analysis set (FAS) who have evaluable PK concentration data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
ratio | 1.33 (0.530) | 1.85 (1.17) | 1.64 (1.41)

10. Secondary Outcome: Change of Tumor Volume From Baseline
Description: This shows the change in tumor volume from baseline to month 6 and from baseline to month 12 in patients treated with pasireotide LAR.
Time Frame: Baseline, Months 6 , 12
Population: FAS: Comprises all patients to whom study treatment has been assigned by randomization. Protocol allowed to change treatment dose (eg, 20mg -> 40mg ->20mg -> 40mg ->60mg) based on efficacy and safety after 3month treatment. So we combined Arms/groups.
Measure: Median (Full Range); unit: mm^3
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
mm^3
  Change from baseline @ Month 6 | -21.0 [-6532.0 to 1002.0]
  Change from baseline @ Month 12 | -1.00 [-4084.0 to 1085.0]

11. Secondary Outcome: Change in Mean GH Levels From Baseline
Description: This shows the change in mean GH levels from baseline in median GH levels by visit.
Time Frame: Baseline, Months 2.75, 3, 6, 9, 12, 18, 24
Population: as for outcome 10
Measure: Median (Full Range); unit: ug/L
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
ug/L
  Change from baseline @ Month 2.75 | -7.60 [-157.2 to 39.3]
  Change from baseline @ Month 3 | -5.98 [-99.2 to 39.3]
  Change from baseline @ Month 6 | -7.27 [-149.8 to 39.3]
  Change from baseline @ Month 9 | -8.83 [-163.8 to 39.3]
  Change from baseline @ Month 12 | -8.90 [-159.2 to 3.0]
  Change from baseline @ Month 18 | -15.68 [-23.9 to 39.3]
  Change from baseline @ Month 24 | -16.67 [-25.5 to -1.4]

12. Secondary Outcome: Change in Ring Size From Baseline
Description: Change of clinical signs from baseline: ring size. In Japan, ring sizes are specified using a numerical scale, that only has whole sizes, and does not have simple linear correlation with diameter or circumference. Only numbers are used ranging from 1 to 27. For instance, a ring size of 1 in Japan is equivalent to an inside circumference ring size of 38.86 mm and a ring size of 27 in Japan is equivalent to an inside circumference ring size of 70.15 mm.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 10
Measure: Median (Full Range); unit: other - Japanese ring size number
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
other - Japanese ring size number
  Month 3 | -1.00 [-3.0 to 0.0]
  Month 6 | -2.00 [-6.0 to 2.0]
  Month 9 | -2.00 [-6.0 to 1.0]
  Month 12 | -2.00 [-6.0 to 1.0]

13. Secondary Outcome: Number of Participants With Acromegaly Symptoms or Pituitary Gigantism (Core Phase)
Description: Number of participants with a change of clinical signs from baseline (BL): headache (HA), fatigue (FA), perspiration (PE), paresthesias (PA), osteoarthralgia (OS)
Time Frame: 12 Months (Core phase)
Population: Full analysis set (FAS) comprises all patients to whom study treatment has been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the study treatment they have been assigned to during the randomization procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg
Number analyzed (Participants) | 11 | 11 | 11
Participants
  HA @ BL: non/absent | 9 | 6 | 10
  HA @ BL: mild | 1 | 4 | 0
  HA @ BL: moderate | 1 | 0 | 0
  HA @ BL: severe | 0 | 0 | 1
  HA @ BL: very severe | 0 | 1 | 0
  HA @ BL: total (all categories) | 11 | 11 | 11
  HA @ most extreme post-BL: total non/absent | 8 | 8 | 7
  HA @ most extreme post-BL: total mild | 3 | 2 | 3
  HA @ most extreme post-BL: total moderate | 0 | 0 | 1
  HA @ most extreme post-BL: total severe | 0 | 1 | 0
  HA @ most extreme post-BL: total very severe | 0 | 0 | 0
  HA @ most extreme post-BL: total (all categories) | 11 | 11 | 11
  FA @ BL: non/absent | 7 | 5 | 6
  FA @ BL: mild | 3 | 3 | 2
  FA @ BL: moderate | 1 | 2 | 3
  FA @ BL: severe | 0 | 1 | 0
  FA @ BL: very severe | 0 | 0 | 0
  FA @ BL: total (all categories) | 11 | 11 | 11
  FA @ most extreme post-BL: total non/absent | 4 | 3 | 5
  FA @ most extreme post-BL: total mild | 4 | 5 | 4
  FA @ most extreme post-BL: total moderate | 3 | 3 | 1
  FA @ most extreme post-BL: total severe | 0 | 0 | 1
  FA @ most extreme post-BL: total very severe | 0 | 0 | 0
  FA @ most extreme post-BL: total (all categories) | 11 | 11 | 11
  PE @ BL: non/absent | 6 | 6 | 3
  PE @ BL: mild | 5 | 3 | 6
  PE @ BL: moderate | 0 | 2 | 2
  PE @ BL: severe | 0 | 0 | 0
  PE @ BL: very severe | 0 | 0 | 0
  PE @ BL: total (all categories) | 11 | 11 | 11
  PE @ most extreme post-BL: total non/absent | 5 | 7 | 7
  PE @ most extreme post-BL: total mild | 5 | 2 | 3
  PE @ most extreme post-BL: total moderate | 1 | 1 | 0
  PE @ most extreme post-BL: total severe | 0 | 1 | 1
  PE @ most extreme post-BL: total very severe | 0 | 0 | 0
  PE @ most extreme post-BL: total (all categories) | 11 | 11 | 11
  OS @ BL: non/absent | 9 | 5 | 7
  OS @ BL: mild | 1 | 1 | 3
  OS @ BL: moderate | 1 | 2 | 1
  OS @ BL: severe | 0 | 2 | 0
  OS @ BL: very severe | 0 | 1 | 0
  OS @ BL: total (all categories) | 11 | 11 | 11
  OS @ most extreme post-BL: total non/absent | 8 | 5 | 6
  OS @ most extreme post-BL: total mild | 1 | 2 | 3
  OS @ most extreme post-BL: total moderate | 2 | 2 | 1
  OS @ most extreme post-BL: total severe | 0 | 1 | 1
  OS @ most extreme post-BL: total very severe | 0 | 1 | 0
  OS @ most extreme post-BL: total (all categories) | 11 | 11 | 11
  PA @ BL: non/absent | 9 | 11 | 9
  PA @ BL: mild | 2 | 0 | 1
  PA @ BL: moderate | 0 | 0 | 1
  PA @ BL: severe | 0 | 0 | 0
  PA @ BL: very severe | 0 | 0 | 0
  PA @ BL: total (all categories) | 11 | 11 | 11
  PA @ most extreme post-BL: total non/absent | 7 | 9 | 9
  PA @ most extreme post-BL: total mild | 4 | 1 | 1
  PA @ most extreme post-BL: total moderate | 0 | 1 | 1
  PA @ most extreme post-BL: total severe | 0 | 0 | 0
  PA @ most extreme post-BL: total very severe | 0 | 0 | 0
  PA @ most extreme post-BL: total (all categories) | 11 | 11 | 11

14. Secondary Outcome: Change From Baseline in Prolactin
Description: Change in prolactin levels from baseline
Time Frame: Baseline, Months 3, 6, 9, 12
Population: as for outcome 10
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
pmol/L
  Month 3 | -43.00 [-609.00 to 1087.00]
  Month 6 | 0.00 [-435.00 to 217.00]
  Month 9 | 0.00 [-479.00 to 913.00]
  Month 12 | 0.00 [-653.00 to 217.00]

15. Secondary Outcome: Total-group Response Rate by Visit (Extension Phase)
Description: Percentage of participants with a reduction of mean GH levels to < 2.5 µg/L and the normalization of IGF-1 to within normal limits (age and sex related) a18 and 24 months of study treatment.
Time Frame: Months 18, 24
Population: FAS: Comprises all patients to whom study treatment has been assigned by randomization. The protocol allowed frequent dose changes even extension phase. In this case, separate data is not meaningful.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants
  Month 18: number analyzed (Participants) | 24
  Month 18 | 12.5 [2.7 to 32.4]
  Month 24: number analyzed (Participants) | 23
  Month 24 | 30.4 [13.2 to 52.9]

16. Secondary Outcome: Percentage of Overall Participants With the Reduction of Mean GH Levels to <2.5 ug/L by Visit (Extension Phase)
Description: Percentage of participants with a reduction of mean GH levels to < 2.5µg/L at 18 and 24 months of study treatment
Time Frame: Months 18, 24
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants
  Month 18: number analyzed (Participants) | 24
  Month 18 | 41.7 [22.1 to 63.4]
  Month 24: number analyzed (Participants) | 23
  Month 24 | 60.9 [38.5 to 80.3]

17. Secondary Outcome: Percentage of Overall Participants With the Normalization of IGF-1 by Visit (Extension Phase)
Description: Percentage of participants with the normalization of IGF-1 to within normal limits (age and sex related) at 18 and 24 months of study. treatment
Time Frame: Months 18, 24
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pasireotide LAR - All Participants
Number analyzed (Participants) | 33
Percentage of participants
  Month 18: number analyzed (Participants) | 24
  Month 18 | 16.7 [4.7 to 37.4]
  Month 24: number analyzed (Participants) | 23
  Month 24 | 30.4 [13.2 to 52.9]

18. Secondary Outcome: Change From Baseline in Mean GH by Visit and SSA Uncontrolled Status (Extension Phase)
Description: This shows a change of mean GH levels and somatostatin analogues (SSAs) from baseline in extension phase
Time Frame: Baselnine, Months 2.75, 3, 6, 9, 12, 18, 24
Population: as for outcome 2
Measure: Median (Full Range); unit: ug/L
Groups:
- SSA Uncontrolled: Somatostatin analogue (SSA) uncontrolled population composes of patients who were pre-treated with SSA for >= 12 weeks.
- Others: Patients who were pre-treated with SSA for < 12 weeks or were not pre-treated with SSA are considered as others.
Arm/Group | SSA Uncontrolled | Others
Number analyzed (Participants) | 20 | 13
ug/L
  Month 2.75 | -8.84 [-25.6 to 39.3] | -6.62 [-157.2 to -1.4]
  Month 3 | -6.71 [-22.2 to 39.3] | -5.04 [-99.2 to -1.4]
  Month 6 | -8.15 [-25.4 to 39.3] | -6.35 [-149.8 to -1.4]
  Month 9 | -9.02 [-24.6 to 39.3] | -8.72 [-163.8 to 1.8]
  Month 12 | -10.10 [-29.1 to 3.0] | -7.29 [-159.2 to -1.4]
  Month 18 | -8.88 [-23.9 to 39.3] | -7.70 [-155.7 to -0.3]
  Month 24 | -9.76 [-25.5 to 39.3] | -6.80 [-32.8 to -1.4]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 1513 days.
Description: Protocol allowed dose modification after month 3 and so analyzing AE separately was did not provide a clinically meaningful data.
Groups:
- Pasireotide LAR - All Participants (All Patieents): Patients who were randomized to the study - regardless of whether they were in the Core or Extension phase.
Arm/Group | Pasireotide LAR 20mg | Pasireotide LAR 40mg | Pasireotide LAR 60mg | Pasireotide LAR - All Participants (All Patieents)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/11 | 5/11 | 11/33
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11 | 11/11 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR 20mg (N=11) | Pasireotide LAR 40mg (N=11) | Pasireotide LAR 60mg (N=11) | Pasireotide LAR - All Participants (All Patieents) (N=33)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR 20mg (N=11) | Pasireotide LAR 40mg (N=11) | Pasireotide LAR 60mg (N=11) | Pasireotide LAR - All Participants (All Patieents) (N=33)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Eustachian tube patulous (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 1
Arteriosclerotic retinopathy (Eye disorders) | 0 | 0 | 1 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1 | 1
Eye discharge (Eye disorders) | 1 | 0 | 0 | 1
Pterygium (Eye disorders) | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal symptom (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3 | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 6
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 3 | 5
Pancreatic duct dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Fatigue (General disorders) | 0 | 2 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 2 | 1 | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 3 | 6
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 0 | 2 | 2
Gallbladder polyp (Hepatobiliary disorders) | 1 | 1 | 1 | 3
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 2 | 0 | 1 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 2
Influenza (Infections and infestations) | 1 | 2 | 0 | 3
Nasopharyngitis (Infections and infestations) | 7 | 6 | 8 | 21
Paronychia (Infections and infestations) | 1 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Venomous sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 2
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 0 | 2
Blood uric acid increased (Investigations) | 0 | 1 | 1 | 2
Blood urine present (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 3 | 3
Insulin-like growth factor decreased (Investigations) | 0 | 1 | 1 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2 | 2 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 2 | 2 | 4
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4 | 4 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cervical polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 4
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
After the first 3 months, pasireotide LAR dose could be increased for efficacy or decreased for safety at any time during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT01673646/SAP_000.pdf
  • Study Protocol (2014-07-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT01673646/Prot_001.pdf